CLINICAL TRIAL: NCT02221817
Title: Prospective, Randomized Trial of Ultrasound Guided and Blind Corticosteroid Injection for Trochanteric Bursitis
Brief Title: Comparison of Ultrasound Guided Versus Blind Corticosteroid Injection for Trochanteric Bursitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1407358564
Record Dates: First submitted 2014-08-16; First posted 2014-08-20 (Estimated); Results first posted 2021-01-20 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-09

CONDITIONS: Bursitis
MeSH Terms: conditions — Bursitis | interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blind (Active Comparator): Trochanter injection
  Interventions: Procedure: Trochanter bursa injections
- Ultrasound (Experimental): Trochanter injection
  Interventions: Procedure: Trochanter bursa injections; Device: Ultrasound

INTERVENTIONS:
Procedure: Trochanter bursa injections
Device: Ultrasound
  Arms: Ultrasound

SUMMARY:
Trochanteric bursitis is a common condition, effecting 20% of the population. \Most with trochanteric bursitis experience chronic intermittent or continuous hip pain at and around the greater trochanter.

The cause of trochanteric bursitis is believed to be a result of inflammation of the bursa, though this has not been confirmed. Accordingly, the use of corticosteroid injections has been shown to provide considerable relief. However, routine "blind" injections, those performed without the aid of imaging, such as fluoroscopy, have shown limited success in the appropriate needle placement. Fortunately, blind injections have yielded positive results in majority of the cases. Additionally, the use of fluoroscopy has not shown to improve clinical outcome for trochanter bursa injections.

Although the use of fluoroscopy has not shown positive benefit, other modes of imaging, such as ultrasound have not been studied and may be more useful. Fluoroscopy allows for bony-landmark based injections. Ultrasound allows for direct visualization of the soft tissue structures such as the bursa and has gained significant support for use in musculoskeletal injections. This prospective blinded study's aim is to evaluate, if any, the benefit of an ultrasound guided injection and whether ultrasound should be routinely used during trochanter bursa injections.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of trochanteric bursitis
2. 18 years of age or older when written informed consent is obtained
3. Signed Institutional Review Board (IRB) approved informed consent form

Exclusion Criteria:

1. Allergy to triamcinolone or bupivicaine
2. Coagulopathy
3. Active Infection
4. Currently diagnosed with cognitive impairment, or exhibits any characteristic, that would limit study candidate's ability to assess pain relief or complete study assessments

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-08; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- West Virginia University Hospitals, Morgantown, West Virginia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was ended and the PI has left the institution. The numbers presented are what was initially entered by the research team. From data available, 80 participants were enrolled on the study; no information about those participants could be located. No other data could be located and it cannot be determined which arm the 80 participants were enrolled in or if they completed the study.
Groups:
- Blind: Trochanter injection
  Trochanter bursa injections
- Ultrasound: Trochanter injection
  Trochanter bursa injections
  Ultrasound
Period: Overall Study
Arm/Group | Blind | Ultrasound
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study was ended and the PI has left the institution. No results information is available, all efforts were to made to retrieve results information, but were unsuccessful. No study data is available.
Groups:
- Total: Total of all reporting groups
Arm/Group | Blind | Ultrasound | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity Measured on Visual Analog Scale (VAS)
Time Frame: 3 month
Population: as for baseline characteristics
Arm/Group | Blind | Ultrasound
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Disability Measured on Becks Disability Scale
Time Frame: Baseline, 2 weeks, 3 month
Population: as for baseline characteristics
Arm/Group | Blind | Ultrasound
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Adverse Effects
Time Frame: 2 weeks, 3 month
Population: as for baseline characteristics
Arm/Group | Blind | Ultrasound
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Pain Improvement
Description: Percent improvement
Time Frame: 2 weeks, 3 months
Population: as for baseline characteristics
Arm/Group | Blind | Ultrasound
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The study was ended and the PI has left the institution. No results information is available, all efforts were to made to retrieve results information, but were unsuccessful. No study data is available.
Arm/Group | Blind | Ultrasound
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This study is considered to be completed, because before leaving the institution the PI indicated the study status as completed and entered that actual enrollment number of 80 participants. No other information could be located or obtained for the study and therefore no specific results information can be included. The study status as completed and actual enrollment number of 80 participants should be considered an accurate representation of all available study information.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes